CLINICAL TRIAL: NCT01111435
Title: A Prospective Study of Spasticity in Individuals With Multiple Sclerosis in Transition From Interferon to Glatiramer Acetate (Copaxone®)
Brief Title: A Prospective Study of Spasticity in Individuals With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fraser, Cira, Ph.D., RN, ACNS-BC (Individual)
Responsible Party: Principal Investigator, Cira Fraser PhD, RN, ACNS-BC, Associate Professor, Fraser, Cira, Ph.D., RN, ACNS-BC
Other Study IDs: Spasticity2010
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with Multiple Sclerosis

SUMMARY:
This study is expected to contribute to the body of knowledge on the benefits of individuals with MS taking glatiramer acetate (Copaxone®). If patients have less spasticity when taking glatiramer acetate (Copaxone®), they may be more likely to have an improved quality of life.

The hypotheses for this study are:

1. Study participants who transition from interferon therapy to glatiramer acetate (Copaxone®) for a six month period will have a decrease in spasticity.
2. Study participants who transition from interferon therapy to glatiramer acetate (Copaxone®) for a six month period will have a change in perceptions of the impact of spasticity on their lives.

DETAILED DESCRIPTION:
The purpose of this study is to determine if there is a change in spasticity and perceptions of the impact of spasticity in individuals with multiple sclerosis who transition from interferon to glatiramer acetate (Copaxone®).•

* Potential participants meeting the criteria will be identified by Shared Solutions and informed of the study. Interested individuals will contact the investigator either by email or telephone. Enrollment will continue until there are 110 participants starting glatiramer acetate (Copaxone®).
* Potential participants will be informed of the details of the study, eligibility will be confirmed, and participant's questions answered.
* The two study instruments and the sociodemographic questionnaire will be emailed or mailed via UPS along with an information letter. May be returned either via email, fax or UPS mail.
* At month 6 for each participant, the study instruments and sociodemographic questionnaire will be sent a second time and returned to the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Stopped interferon (beta-1a or beta-1b) within the past 30 days
* About to start or started glatiramer acetate (Copaxone®) within the past 21 days.
* At least 18 years of age
* Has spasticity at the beginning of the study
* Able to ambulate with unilateral support or without support
* Understands, speaks and reads English

Exclusion Criteria:

* Severe Gait Disability or Total Gait Disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Multiple Sclerosis living in the community
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Spasticity Scale | Administered at 6 month follow-up

SECONDARY OUTCOMES:
Performance Scales (Measure of Disability) | Administered at 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Cira Fraser, PHD, Principal Investigator — Monmouth University
Locations (1):
- Shared Solutions Call Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Meca-Lallana, J.E., Amorin-Diaz, M., Martinez-Navarro, M.L. & Fernandez- Barreiro, A. (2008). Spasticity in multiple sclerosis: A pilot study to evaluate the efficacy of glatiramer acetate. Multiple Sclerosis, 145 (Suppl. 2), S165.